CLINICAL TRIAL: NCT02691468
Title: Comparison of Displacement Between Polyvinyl Chloride(PVC) and Silicon Double-Lumen Endobronchial Tubes(DLT) During Change of Position
Brief Title: Displacement Between PVC and Silicon DLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Associate Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YeungnamUDLT
Record Dates: First submitted 2016-02-05; First posted 2016-02-25 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure; Surgical Procedure, Unspecified
Keywords: one lung ventilation; double lumen endobronchial tube; displacement; Fiberoptic bronchoscope

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVC DLT (Active Comparator): After the induction of general anesthesia, a left sided PVC DLT was placed by the anesthesiologist using direct laryngoscopy. Tube position was confirmed with fiberotic bronchoscope.
  The first set of measurements tracheal distance(from tracheal carina to proximal tip of DLT) and bronchial distance(from bronchial carina to distal tip of DLT) measured by bronchoscope is taken in supine position .
  The second set of measurements is taken in lateral position after position change.
  The displacement of PVC DLT is calculated from difference in tracheal distance between supine and lateral position.
  Interventions: Device: PVC DLT
- silicon DLT (Active Comparator): After the induction of general anesthesia, a left sided silicon DLT was placed by the anesthesiologist using direct laryngoscopy. Tube position was confirmed with fiberotic bronchoscope.
  The first set of measurements tracheal distance(from tracheal carina to proximal tip of DLT) and bronchial distance(from bronchial carina to distal tip of DLT) measured by bronchoscope is taken in supine position .
  The second set of measurements is taken in lateral position after position change.
  The displacement of silicon DLT is calculated from difference in tracheal distance between supine and lateral position.
  Interventions: Device: silicon DLT

INTERVENTIONS:
Device: PVC DLT — PVC DLT is type of double lumen tube that is composed of PVC
  Other Names: PVC double-lumen tube
  Arms: PVC DLT
Device: silicon DLT — silicon DLT is type of double lumen tube that is composed of silicon
  Other Names: silicon double-lumen tube
  Arms: silicon DLT

SUMMARY:
The purpose of this study is to compare difference of displacement between Polyvinyl Chloride(PVC) and Silicon double-lumen endobronchial tubes(DLTs) during changing position from supine to lateral in thoracic surgery.

DETAILED DESCRIPTION:
Lung isolation and differential lung ventilation, resulting in collapse of operative lung and ventilation of non-operating lung (one lung ventilation; OLV) are essential for thoracic surgery in lung, esophagus and thoracic aorta.

DLT, consisted of tracheal and bronchial lumens, is commonly used to perform differential lung ventilation. The correct position of each lumen in trachea and main bronchus is essential for successful OLV. However, DLT displacement occurs commonly while patients are changed position from the supine to the lateral. The deleterious consequences of a malpositioned DLT can be substantial, even life-threatening including severe hypoxemia.

Considering displacement of DLT during position change and surgical traction, previous studies recommended endobronchial cuff of DLT should be positioned at 0.5cm below the tracheal carina when using left-sided DLT. However, it is based on the data from several research conducted by PVC DLT.

These days, Silicon DLT, different in material from PVC DLT, is also widely used in clinical practice. Silicon DLT is different in not only position of ballon but also distance of each lumen. Furthermore,there are no identified studies about the displacement of silicon DLT during patient position change in thoracic surgery.

Therefore, it is necessary to measure the movement of silicon DLT during positional change from supine to lateral for finding the proper positioning of DLT.

The investigators compare the difference of displacement between PVC DLT and silicon DLT distance during positional change from supine to lateral by fiberotic bronchoscope. And the investigators try to find proper position of PVC and silicon DLT, respectively, to perform safe and successful OLV during thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient required differential lung ventilation in elective thoracic surgery American society of Anesthesiologist physical status(ASA PS) 1~3

Exclusion Criteria:

* emergency surgery, difficult intubation, poor lung function to accomplish OLV during surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee applejsm@gmail.com, MD, Principal Investigator — Yeungnam University College of Medicine
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benumof JL, Partridge BL, Salvatierra C, Keating J. Margin of safety in positioning modern double-lumen endotracheal tubes. Anesthesiology. 1987 Nov;67(5):729-38. doi: 10.1097/00000542-198711000-00018. PMID 3674473
- [Background] Desiderio DP, Burt M, Kolker AC, Fischer ME, Reinsel R, Wilson RS. The effects of endobronchial cuff inflation on double-lumen endobronchial tube movement after lateral decubitus positioning. J Cardiothorac Vasc Anesth. 1997 Aug;11(5):595-8. doi: 10.1016/s1053-0770(97)90011-2. PMID 9263092
- [Background] Yoon TG, Chang HW, Ryu HG, Kwon TD, Bahk JH. Use of a neck brace minimizes double-lumen tube displacement during patient positioning. Can J Anaesth. 2005 Apr;52(4):413-7. doi: 10.1007/BF03016286. PMID 15814758
- See also: Margin of safety in positioning modern double-lumen endotracheal tubes. Anesthesiology. — http://www.ncbi.nlm.nih.gov/pubmed/3674473
- See also: The effects of endobronchial cuff inflation on double-lumen endobronchial tube movement after lateral decubitus positioning. — http://www.ncbi.nlm.nih.gov/pubmed/9263092
- See also: Use of a neck brace minimizes double-lumen tube displacement during patient positioning. — http://www.ncbi.nlm.nih.gov/pubmed/15814758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and eight adult patients, aged between 18 and 75 years, American Society of Anesthesiologists (ASA) physical status 1 ~ 3 scheduled for elective thoracic surgery were enrolled.
Pre-assignment Details: Patients with emergency surgery, difficult intubation, poor lung function to accomplish one-lung ventilation (OLV) during surgery were excluded.
Groups:
- Polyvinyl Chloride (PVC) Double Lumen Tube (DLT): After the induction of general anesthesia, a left sided PVC DLT was placed by the anesthesiologist using direct laryngoscopy. Tube position was confirmed with fiberotic bronchoscope.
  The first set of measurements tracheal distance(from tracheal carina to proximal tip of DLT) and bronchial distance(from bronchial carina to distal tip of DLT) measured by bronchoscope is taken in supine position .
  The second set of measurements is taken in lateral position after position change.
  The displacement of PVC DLT is calculated from difference in tracheal distance between supine and lateral position.
  PVC DLT: PVC DLT is type of double lumen tube that is composed of polyvinlyl chloride.
- Silicon Double Lumen Tube (DLT): After the induction of general anesthesia, a left sided silicon DLT was placed by the anesthesiologist using direct laryngoscopy. Tube position was confirmed with fiberotic bronchoscope.
  The first set of measurements tracheal distance(from tracheal carina to proximal tip of DLT) and bronchial distance(from bronchial carina to distal tip of DLT) measured by bronchoscope is taken in supine position .
  The second set of measurements is taken in lateral position after position change.
  The displacement of silicon DLT is calculated from difference in tracheal distance between supine and lateral position.
  silicon DLT: silicon DLT is type of double lumen tube that is composed of silicon
Period: Overall Study
Arm/Group | Polyvinyl Chloride (PVC) Double Lumen Tube (DLT) | Silicon Double Lumen Tube (DLT)
Started | 54 | 54
Completed | 48 | 52
Not Completed | 6 | 2
Not completed — Bronchial blocker use | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Failure to advance FOB | 2 | 0

BASELINE CHARACTERISTICS:
Population: 108 adult patients scheduled for elective thoracic surgery were enrolled. They were randomly allocated into two groups using a computer-generated random assignment scheme; group P (Polyvinyl chloride (PVC) double lumen tube (DLT)) and group S (Silicone DLT).
Groups:
- PVC DLT: After the induction of general anesthesia, a left sided PVC DLT was placed by the anesthesiologist using direct laryngoscopy. Tube position was confirmed with fiberotic bronchoscope.
  The first set of measurements tracheal distance(from tracheal carina to proximal tip of DLT) and bronchial distance(from bronchial carina to distal tip of DLT) measured by bronchoscope is taken in supine position .
  The second set of measurements is taken in lateral position after position change.
  The displacement of PVC DLT is calculated from difference in tracheal distance between supine and lateral position.
  PVC DLT: PVC DLT is type of double lumen tube that is composed of PVC
- Silicon DLT: After the induction of general anesthesia, a left sided silicon DLT was placed by the anesthesiologist using direct laryngoscopy. Tube position was confirmed with fiberotic bronchoscope.
  The first set of measurements tracheal distance(from tracheal carina to proximal tip of DLT) and bronchial distance(from bronchial carina to distal tip of DLT) measured by bronchoscope is taken in supine position .
  The second set of measurements is taken in lateral position after position change.
  The displacement of silicon DLT is calculated from difference in tracheal distance between supine and lateral position.
  silicon DLT: silicon DLT is type of double lumen tube that is composed of silicon
- Total: Total of all reporting groups
Arm/Group | PVC DLT | Silicon DLT | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants] — Population: inclusion in final analysis
  Participants
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 20 | 47 | 67
    >=65 years | 33 | 7 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (16.1) | 57.8 (14.9) | 57.3 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: inclusion in final analysis
  Participants
    Female | 18 | 18 | 36
    Male | 36 | 36 | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: the Incidence of Clinically Significant Displacement of DLTs During Change of Patient Position
Description: The tracheal distance was defined as the distance between the distal tip of the tracheal lumen and tracheal carina whereas the bronchial distance was defined as that between the bronchial carina and distal tip of endobronchial lumen. The displacement of DLT was determined by changes in tracheal and bronchial distances, obtained by subtracting supine measurements from lateral measurements and subtracting measurements at start of surgery from measurements at the end of surgery, respectively. Clinically significant displacement was defined when the DLT was deviated by more than 10 mm from the initial correct position, regardless of the direction of displacement.
Time Frame: from supine to lateral decubitus position during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | PVC DLT | Silicon DLT
Number analyzed (Participants) | 48 | 52
Participants | 17 | 18

2. Secondary Outcome: the Incidence of Critical Malposition of DLTs
Description: The displacement of DLT was determined by changes in tracheal and bronchial distances, obtained by subtracting supine measurements from lateral measurements and subtracting measurements at start of surgery from measurements at the end of surgery, respectively. The critical malposition was defined when the DLT was required repostion for successful OLV during position change
Time Frame: from supine to lateral decubitus position
Measure: Number; unit: participants
Arm/Group | PVC DLT | Silicon DLT
Number analyzed (Participants) | 48 | 52
participants | 4 | 4

ADVERSE EVENTS:
Time Frame: from induction of anesthesia through study completion, an average of 5 hours
Description: Hypoxemia : oxygen saturation less than 93%
Arm/Group | PVC DLT | Silicon DLT
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

LIMITATIONS AND CAVEATS:
First, the position change and surgical manipulation may have a combined. Second, we did not monitor the pressure and volume of air injected into the bronchial cuff. Third, we did not investigate ideal position of DLT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02691468/Prot_SAP_000.pdf